CLINICAL TRIAL: NCT04798768
Title: Effectiveness of the EMPOWER™ Modular Pacing System and EMBLEM™ Subcutaneous ICD to Communicate Antitachycardia Pacing
Acronym: MODULAR ATP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1907
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Tachycardia, Ventricular; Arrhythmia, Ventricular
MeSH Terms: conditions — Tachycardia, Ventricular; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MODULAR ATP Study Participants (Experimental): All subjects that signed the informed consent were included.
  Patients consented to receive the mCRM Therapy System which consists of the EMPOWER Leadless Pacemaker and an EMBLEM S-ICD upgraded with investigational firmware.
  Interventions: Device: mCRM Therapy System

INTERVENTIONS:
Device: mCRM Therapy System — Communication testing between S-ICD and LCP in 4 body postures as well as required electrical testing.
  Other Names: Communication of S-ICD to Leadless Cardiac Pacemaker (LCP)

SUMMARY:
The MODULAR ATP Clinical Study is designed to demonstrate safety, performance, and effectiveness of the Modular Cardiac Rhythm Management (mCRM) Therapy System.

DETAILED DESCRIPTION:
The MODULAR ATP Clinical Study will enroll subjects with a standard Implantable Cardioverter Defibrillator (ICD) indication applying international practice guidelines, as well as those who already have an implanted S-ICD System and satisfy the inclusion criteria for this study, while not meeting any exclusion criteria. Subjects will be followed for at least 6 months following mCRM Therapy System implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient who meets Class I, IIa, or IIb guideline ICD indications[i],[ii], or who has an existing TV-ICD[iii] or S-ICD[iv]
* Patient who is deemed to be at risk for MVT based on at least ONE of the following:

  * History of Non-Sustained MVT with LVEF ≤ 50%
  * History of sustained VT/VF (secondary prevention) with LVEF ≤ 50% or significant cardiac scar*
  * History of syncope deemed to be arrhythmic in origin
  * History of ischemic cardiomyopathy with LVEF ≤35%
  * History of non-ischemic cardiomyopathy with LVEF ≤35% and significant scar*
* Patient who is willing and capable of providing informed consent (which is not to include the use of a legally authorized representative (LAR) for documentation of informed consent) and participating in all testing associated with this investigation at an approved study site and at the intervals defined by this protocol
* Patient who is age 18 years or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Patient with an ongoing complication due to Cardiac Implantable Electronic Device (CIED) infection or CIED explant
* Transvenous lead remnants within the heart from a previously implanted CIED (Note: transvenous lead remnants outside the heart (e.g., in the SVC) are allowed)
* Patient with a known LA thrombus
* Patient with a ventricular arrhythmia due to a reversible cause
* Patient indicated for implantation of a dual chamber pacemaker or cardiac resynchronization therapy (CRT)
* Patient with another implanted medical device that could interfere with implant of the leadless pacemaker, such as an implanted inferior vena cava filter or mechanical tricuspid heart valve
* Patient requires rate-responsive pacing therapy
* Patient is entirely pacemaker-dependent (defined as escape rhythm ≤ 30 bpm)
* Patient with Acute Coronary Syndrome (i.e. Acute Myocardial Infarction, Unstable Angina) within 40 days
* Inability to access femoral vein with a 21-French or larger inner diameter introducer sheath due to known anatomy condition, recent surgery, and/ or other relevant condition
* Patient who has an active implanted electronic medical device intended for chronic use concomitantly with the study system, such as a left ventricular assist device (LVAD). Note that a temporary pacing wire is allowed.
* Patient with known or suspected sensitivity to Dexamethasone Acetate (DXA)
* Patient with a known cardiovascular anatomy that precludes implant in the right ventricle
* Patient with a known allergy to any system components
* Patient with a known or suspected intolerance to S-ICD conversion testing, based on physician discretion
* Patient is not likely to have meaningful survival** for at least 12 months (documented or per investigator's discretion)
* Patient is enrolled in any other concurrent study. Co-enrollment into other studies such as observational studies/ registries needs prior written approval by BSC. Local mandatory governmental registries are accepted for co-enrollment without approval by BSC.
* Patient who is a woman of childbearing potential who is known to be pregnant at the time of study enrollment (method of assessment upon investigator's discretion)

  [i]Al-Khatib, et al. 2017 AHA/ACC/HRS Guideline for Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death. A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Circulation. (2018); 138:e272-e391.

[ii] 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: The Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC). European Heart Journal (2015) 36, 2793-2867.

[iii] TV-ICD system is expected to be fully explanted during or prior to full Coordinated System implant

[iv] Potential subjects with a Model 1010 S-ICD Pulse Generator are only eligible for MODULAR ATP if they are getting upgraded to Model A209, A219 or future BSC S-ICD Pulse Generator; Patients with an existing S-ICD PG subject to the electrical overstress field action are only eligible for MODULAR ATP if they are getting a new BSC Model A209 or A219, or future BSC S-ICD Pulse Generator

*Significant cardiac scar is defined as a scar involving at least one ventricular myocardial segment (i.e., basal infero-septum) as identified in the official findings of a cMRI, or nuclear viability study, or echo report by the interpreting radiologist/ cardiologist who is not affiliated with the study

**meaningful survival means that a patient has a reasonable quality of life and functional status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2030-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lloyd, MD, Principal Investigator — Emory University; Reinoud Knops, MD, PhD, Principal Investigator — Amsterdam University Medical Centre; Lluis Mont, MD, PhD, Principal Investigator — Hospital Clinic, University of Barcelona; Vivek Reddy, MD, Principal Investigator — The Mount Sinai Hospital
Locations (38):
- United States (18):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - AdventHealth Orlando, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Baptist Health Lexington, Lexington, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Cooper Hospital - University Medical Center, Camden, New Jersey
  - Northwell University Hospital, Manhasset, New York
  - Mount Sinai Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Sentara Norfolk General, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Kepler Universitaetsklinikum, Linz, Austria
- Canada (2):
  - Institut de Cardiologie de Quebec (Montreal Heart), Montreal, Quebec
  - Institut Universitaire de Cardilogie et Pnuemologie de Quebec (IUCPQ), Québec
- Na Homolce Hospital, Prague, Czechia
- France (4):
  - CHU Grenoble - Hospital Michallon, Grenoble
  - CHRU de Lille, Lille
  - CHU de Nantes-Hopital Laennec, Nantes
  - Hospital European Georges-Pompidou, Paris
- Italy (4):
  - Spedali Civil di Brescia, Brescia
  - Maria Cecilia Hospital SPA, Cotignola
  - AZ Osp Monaldi, Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Netherlands (3):
  - Amsterdam University Medical Center, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC University Medical Center, Rotterdam
- Hospital Clinic of Barcelona, Barcelona, Spain
- United Kingdom (4):
  - The General Infirmary, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - Manchester Heart Center, Manchester
  - Southampton University Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers in this study.

REFERENCES:
- [Background] Lloyd MS, Brisben AJ, Reddy VY, Blomstrom-Lundqvist C, Boersma LVA, Bongiorni MG, Burke MC, Cantillon DJ, Doshi R, Friedman PA, Gras D, Kutalek SP, Neuzil P, Roberts PR, Wright DJ, Appl U, West J, Carter N, Stein KM, Mont L, Knops RE. Design and rationale of the MODULAR ATP global clinical trial: A novel intercommunicative leadless pacing system and the subcutaneous implantable cardioverter-defibrillator. Heart Rhythm O2. 2023 Jun 2;4(7):448-456. doi: 10.1016/j.hroo.2023.05.004. eCollection 2023 Jul. PMID 37520021
- [Result] Knops RE, Lloyd MS, Roberts PR, Wright DJ, Boersma LVA, Doshi R, Friedman PA, Neuzil P, Blomstrom-Lundqvist C, Bongiorni MG, Burke MC, Gras D, Kutalek SP, Amin AK, Fu EY, Epstein LM, Tolosana JM, Callahan TD, Aasbo JD, Augostini R, Manyam H, Nair DG, Mondesert B, Su WW, Pepper C, Miller MA, Grammes J, Saleh K, Marquie C, Merchant FM, Cha YM, Cunnington C, Frankel DS, West J, Matznick E, Swackhamer B, Brisben AJ, Weinstock J, Stein KM, Reddy VY, Mont L; MODULAR ATP Investigators. A Modular Communicative Leadless Pacing-Defibrillator System. N Engl J Med. 2024 Oct 17;391(15):1402-1412. doi: 10.1056/NEJMoa2401807. Epub 2024 May 18. PMID 38767244
- [Derived] Lloyd MS, Reddy VY, Roberts P, Doshi RN, Wright DL, Boersma LVA, Friedman PA, Neuzil P, Blomstrom-Lundqvist C, Bongiorni MG, Burke MC, Gras D, Kutalek SP, Marijon E, Tolosana JM, Amin AK, Epstein LM, Aasbo JD, Callahan TD, Brisben AJ, West J, Matznick E, Speakman B, Bachman TN, Mont L, Knops RE. One-Year Outcomes of the MODULAR ATP Trial: A Novel Leadless Pacemaker in Wireless Communication With a Subcutaneous Implantable Cardioverter Defibrillator. Circ Arrhythm Electrophysiol. 2026 Jan;19(1):e014395. doi: 10.1161/CIRCEP.125.014395. Epub 2025 Nov 13. PMID 41231774

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Implanted With S-ICD and Leadless Cardiac Pacemaker: Patients implanted with an S-ICD and leadless cardiac pacemaker that complete intended testing based on the study protocol
  mCRM Therapy System: Communication testing between S-ICD and LCP in 4 body postures as well as required electrical testing.
Period: Overall Study
Arm/Group | Patients Implanted With S-ICD and Leadless Cardiac Pacemaker
Started | 297
Implanted With mCRM Therapy System or Attempt or Partial Implant | 288
Implanted With mCRM Therapy System or Attempt | 287
Implanted With mCRM Therapy System | 286
Interim Analysis Cohort | 162 (Pre-specified interim analysis for 6 month endpoints)
CE Mark Cohort | 117 (Pre-specified 12-month safety analysis for CE Mark submission)
Completed (Study is ongoing. As of the date of the snapshot, 264 subjects are actively being followed) | 0
Not Completed | 297

BASELINE CHARACTERISTICS:
Groups:
- MODULAR ATP Study Participants: Patients consented to receive the mCRM Therapy System which consists of the EMPOWER Leadless Pacemaker and an EMBLEM S-ICD upgraded with investigational firmware
Arm/Group | MODULAR ATP Study Participants
Number analyzed (Participants) | 297
Age, Continuous [Mean (Standard Deviation); unit: Years] — All subjects that signed the study informed consent were included
  Years | 59 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 245
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 177
  Black or African American | 23
  Asian | 6
  American Indian or Alaska native | 2
  Other | 2
  Not disclosed | 76
  Multiracial | 11
Region of Enrollment [Number; unit: participants]
  Canada | 16
  Netherlands | 12
  Austria | 5
  United States | 180
  Czechia | 1
  United Kingdom | 18
  Italy | 15
  France | 30
  Spain | 20
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (6.4)
LVEF [Mean (Standard Deviation); unit: percent] | 35.3 (13.1)
NYHA Classification [Count of Participants; unit: Participants] — NYHA Classification of severity of heart failure places subjects in 1 of 4 categories based on how much they are limited during physical activity, based on physician assessment.
  Class I = normal function status, Class II = Slight limitation of functional status, Class III = Marked limitation of functional status, Class IV = Severe limitation of functional status.
  Participants
    Class I | 88
    Class II | 146
    Class III | 61
    Class IV | 2
Prevention status [Count of Participants; unit: Participants]
  Primary Prevention | 170
  Secondary Prevention | 127
Ischemic cardiomyopathy [Count of Participants; unit: Participants] | 182
Non-ischemic cardiomyopathy [Count of Participants; unit: Participants] | 93
Diabetes [Count of Participants; unit: Participants] | 108
Renal dysfunction [Count of Participants; unit: Participants] | 47
Hyperlipidemia [Count of Participants; unit: Participants] | 181

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint 1: Percentage of Subjects Without Major EMPOWER MPS System- or Procedure-Related Complications Through 6 Months
Description: Major EMPOWER MPS System- and Procedure-related Complication-Free Rate Subjects will be assessed for safety issues related to the procedure or system through 6 months post implant
Time Frame: Implant through 6 Months Post-Implant
Measure: Number (98.8% Confidence Interval); unit: % of subjects free from complication
Groups:
- Interim Analysis Cohort: This subject cohort was determined by the point in time at which 134 subjects (pre-specified in the endpoint design) had a 6 Month Visit with data submitted in the database. Once the 134th subject that fulfilled that requirement was identified, their EMPOWER LP implant date was used to determine the cohort. Any subject with an EMPOWER LP implant or attempted EMPOWER LP implant on or before the identified implant date is included, even if their 6-month follow-up was after the identified subject. This resulted in 162 subjects to be included in the Interim Analysis Cohort.
Arm/Group | Interim Analysis Cohort
Number analyzed (Participants) | 162
% of subjects free from complication | 97.5 [92.5 to NA] — One-sided test was performed with 1.2% alpha. Lower one-sided 98.8% confidence limit was compared to performance goal of 86%. It was pre-specified to only calculate the lower confidence interval.

2. Primary Outcome: Safety Endpoint 2: Percentage of Subjects Without Major EMPOWER MPS System- or Procedure-Related Complications Through 12 Months
Description: Major EMPOWER MPS System- and Procedure-related Complication-free Rate
  Subjects will be assessed for safety issues related to the procedure or system through 12 months post implant
Time Frame: Implant through 12 Months Post-Implant
Measure: Number (97.5% Confidence Interval); unit: % of subjects free from complication
Groups:
- CE Mark Cohort: This subject cohort was determined by the point in time at which 112 subjects had a 12 Month Visit with data submitted in the database. Once the 112th subject that fulfilled that requirement was identified, their EMPOWER LP implant date was used to determine the cohort. Any subject with an EMPOWER LP implant or attempted EMPOWER LP implant on or before the determined implant date is included, even if their 12 Month Visit occurred after subject the identified subject. This resulted in 117 subjects to be included in the CE Mark Analysis Cohort.
Arm/Group | CE Mark Cohort
Number analyzed (Participants) | 117
% of subjects free from complication | 98.3 [93.3 to NA] — One-sided test was performed with 2.5% alpha. Lower one-sided 97.5% confidence limit was compared to performance goal of 81%. It was pre-specified to only calculate the lower confidence interval.

3. Primary Outcome: Primary Effectiveness Endpoint 1: Percentage of Body Postures With Communication Success Between the S-ICD and EMPOWER PG
Description: Communication Success between the S-ICD and EMPOWER PG
  Data from subjects will be assessed for effectiveness of communication between S-ICD and the EMPOWER PG by evaluating if a paced beat is present during communication testing in four postures: upright, supine, and right and left side.
Time Frame: At the 6 Month Follow-up
Population: Number of subjects in the interim analysis cohort who underwent S-ICD to EMPOWER LP communication testing at 6 months in at least one of four postures. Results were adjusted using a repeated measures logistic regression model
Measure: Number (97.5% Confidence Interval); unit: Adjusted % with successful communication
Units Other Than Participants: Postures
Arm/Group | Interim Analysis Cohort
Number analyzed (Participants) | 149
Number analyzed (Postures) | 589
Adjusted % with successful communication | 98.8 [97.0 to NA] — One-sided test was performed with 2.5% alpha. Lower one-sided 97.5% confidence limit was compared to performance goal of 88%. It was pre-specified to only calculate the lower confidence interval.

4. Primary Outcome: Primary Effectiveness Endpoint 2: Percentage of Subjects Classified as a Pacing Capture Threshold (PCT) Responder
Description: Proportion of Subjects with Adequate Pacing Capture Threshold
  Effectiveness will be confirmed by evaluating the percentage of subjects considered to be a PCT Responder, defined as a subject with a PCT measurement of ≤ 2.0 V @ 0.4 ms pulse width
Time Frame: At the 6 Month Follow-up
Population: Number of subjects in the interim analysis cohort with Pacing Capture Threshold data at 6 months
Measure: Number (97.5% Confidence Interval); unit: % of subjects with PCT <= 2V @ 0.4 ms
Arm/Group | Interim Analysis Cohort
Number analyzed (Participants) | 151
% of subjects with PCT <= 2V @ 0.4 ms | 97.4 [93.4 to NA] — One-sided test was performed with 2.5% alpha. Lower one-sided 97.5% confidence limit was compared to performance goal of 80%. It was pre-specified to only calculate the lower confidence interval.

5. Secondary Outcome: Secondary Effectiveness Endpoint: Subject-specific Slope of EMPOWER PG Sensor-Indicated Rate to the Subject's Workload on Treadmill Test
Description: Metabolic-Chronotropic Relation Slope (MCR Slope) from the Kay-Wilkoff Model
  Using the Kay-Wilkoff model, data will be assessed to evaluate the proportionality of the EMPOWER PG's sensor-indicated rate to the subject's workload during the treadmill test
Time Frame: At the 3 Month Visit
Population: Data for this endpoint were obtained from the subset of subjects who consented into the substudy and performed treadmill testing at 3 months
Measure: Mean (95% Confidence Interval); unit: Beta coefficient
Arm/Group | Patients Implanted With S-ICD and Leadless Cardiac Pacemaker
Number analyzed (Participants) | 35
Beta coefficient | 0.96 [0.91 to 1.02]

6. Secondary Outcome: Secondary Safety Endpoint
Description: All-Cause Survival; data not reported as it is still being collected
Time Frame: Implant through 2 years post-implant
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: Entire available follow up: implant through 3.5 years to-date (median participant follow up = 1.3 years)
Description: Adverse event data includes Serious/ non-serious, related/ unrelated to device were to be reported to Boston Scientific by investigational sites. All-cause mortality evaluated in all enrolled subjects (N=297). Adverse Events were evaluated in subjects implanted or attempted with S-ICD and/ or EMPOWER Leadless Pacemaker (N=288).
Groups:
- MODULAR ATP Study Participants: All-cause mortality evaluated in all enrolled participants (N=297). Adverse events were evaluated for participants implanted or attempted with the mCRM Therapy System (S-ICD after study enrollment, and/ or the EMPOWER LP), N=288. Individual adverse event categories evaluated in participants at risk for that event category (287 Leadless Cardiac Pacemaker, 9 TV Lead Extraction Procedure, 288 remaining adverse event categories).
Arm/Group | MODULAR ATP Study Participants
All-Cause Mortality (participants affected / at risk) | 18/297
Serious Adverse Events (participants affected / at risk) | 113/288
Other Adverse Events (participants affected / at risk) | 86/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MODULAR ATP Study Participants (N=288)
Non-cardiovascular (Blood and lymphatic system disorders) | 1 (1)
Cardiovascular (Cardiac disorders) | 54 (86)
Non-cardiovascular (Endocrine disorders) | 6 (7)
Non-cardiovascular (Gastrointestinal disorders) | 5 (6)
Cardiovascular (General disorders) | 7 (9)
Non-cardiovascular (General disorders) | 10 (13)
Non-cardiovascular (Infections and infestations) | 13 (17)
Leadless Cardiac Pacemaker - Procedure (Injury, poisoning and procedural complications) | 13/287 (16)
S-ICD Defibrillation and Conversion Testing (Injury, poisoning and procedural complications) | 2 (3)
S-ICD System Patient Related (Injury, poisoning and procedural complications) | 2 (2)
S-ICD System Procedure (Injury, poisoning and procedural complications) | 7 (8)
TV Lead Extraction Procedure (Injury, poisoning and procedural complications) | 2/9 (4)
Non-cardiovascular (Nervous system disorders) | 2 (2)
Leadless Cardiac Pacemaker - Right Ventricle - Brady (Product Issues) | 1/287 (1)
Modular System (LCP+S-ICD) (Product Issues) | 2 (2)
S-ICD Electrode (Product Issues) | 3 (3)
S-ICD PG (Product Issues) | 2 (2)
S-ICD System Diagnosis (Product Issues) | 2 (2)
S-ICD System Therapy (Product Issues) | 9 (9)
Non-cardiovascular (Renal and urinary disorders) | 9 (12)
Non-cardiovascular (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Non-cardiovascular (Skin and subcutaneous tissue disorders) | 2 (2)
Cardiovascular (Vascular disorders) | 16 (17)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MODULAR ATP Study Participants (N=288)
Cardiovascular (Cardiac disorders) | 25 (29)
Non-cardiovascular (Endocrine disorders) | 1 (1)
Non-cardiovascular (Gastrointestinal disorders) | 1 (1)
Cardiovascular (General disorders) | 8 (9)
Non-cardiovascular (General disorders) | 4 (4)
S-ICD System Patient Related (General disorders) | 2 (2)
Non-cardiovascular (Infections and infestations) | 1 (1)
Leadless Cardiac Pacemaker - Procedure (Injury, poisoning and procedural complications) | 12/287 (12)
Leadless Cardiac Pacemaker - Right Ventricle - Brady (Injury, poisoning and procedural complications) | 1/287 (1)
S-ICD Defibrillation and Conversion Testing (Injury, poisoning and procedural complications) | 1 (1)
S-ICD System Patient Related (Injury, poisoning and procedural complications) | 2 (2)
S-ICD System Procedure (Injury, poisoning and procedural complications) | 16 (18)
Non-cardiovascular (Musculoskeletal and connective tissue disorders) | 1 (1)
Modular System (LCP+S-ICD) (Product Issues) | 2 (2)
S-ICD Electrode (Product Issues) | 1 (1)
S-ICD PG (Product Issues) | 2 (2)
S-ICD System Therapy (Product Issues) | 9 (10)
Cardiovascular (Vascular disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
The study is limited by the nonrandomized design with no comparator group. Prespecified goals for safety and performance were used to define endpoints. Patients were selected with a high risk of ventricular tachycardia. The findings may not be generalizable to other patients who require S-ICDs or who have S-ICDs already implanted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit publication to Sponsor for review at least 60 days prior to submission. Sponsor reserves the right to delete any confidential info or other proprietary info of Sponsor (not incl. Results). Sponsor may extend 90 days to protect its intellectual property (IP) interests. PI shall be free to publish the results of the study after: Initial Publication is published; notification by Sponsor that Initial Publication is no longer planned; or 12 mo. after the expiration date at all sites

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT04798768/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT04798768/SAP_002.pdf